CLINICAL TRIAL: NCT05328063
Title: Impact of Manual Therapy on the Coxofemoral Joint in Patients With Chronic Low Back Pain of Non-Specific Origin.
Brief Title: Is Hip Range of Motion Relevant in the Treatment of Chronic Low Back Pain?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/2022/1/002
Record Dates: First submitted 2022-03-30; First posted 2022-04-14 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-03

CONDITIONS: Chronic Low-back Pain
Keywords: Hip Joint; Gluteus Maximus; Manual Therapy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group. Gluteus maximus strengthening specific program (Experimental)
  Interventions: Other: Control group
- Intervention group. Specific manual therapy program for hip joint and Gluteus maximus strengthening (Experimental)
  Interventions: Other: Control group; Other: Intervention group

INTERVENTIONS:
Other: Control group — All subjects will carry out a gluteus maximus strengthening work out. The exercises should be performed at a frequency of 3 times/week and with a dosage of 3 sets of 8 repetitions.
  1-4 Weeks: 1. Bilateral gluteal bridge: Supine decubitus with knees and hips bent and feet supported. To raise the pelvis until the knees are flexed to 90° and then returns to the starting position. 2.Clam shell: Lateral decubitus with knees and hips bent to 45º, working leg placed on top of the other. Separate this knee while feet remain in contact using a medium density Theraband on the distal thighs. Bilateral work. 3. Side-Step: Bipedestation with Knees and hips bent. The exercise then consists of two steps taken in one direction followed by two steps in the opposite direction to return to the starting position. The elastic band shall be placed above the knees.
  4-8 Weeks: 1.Unilateral gluteal bridge. 2 Clam shell: hips bents to 60º. 3. Side-Step: placing the elastic band over the ankles
Other: Intervention group — All subjects will receive a specific program of manual therapy on the hip joint. 10 sessions of manual therapy will be applied during 8 weeks, 1 session per week, except the first week when two sessions will be applied.
  The protocol consists of passive manual joint therapy at low speed on the hip, applying each mobilization in 3 series of 10 repetitions. It also includes muscle stretching, performing 3 series and holding the stretch for 25 seconds.
  Manual therapy includes: 1. Anteroposterior (AP) and posteroanterior (PA) displacement of the hip. 2. Lateromedial and mediolateral displacement of the hip. 3. Distraction of the long axis/traction of the hip. 4. Lower slip in internal rotation (IR) and external rotation (ER) of the hip. 5. Iliopsoas stretch. 6. Piriformis stretch.To perform the protocol, the patient shall be placed in the supine decubitus position.
  In addition to the same gluteus maximus strengthening programme used for the control group.
  Arms: Intervention group. Specific manual therapy program for hip joint and Gluteus maximus strengthening

SUMMARY:
The study will be carried out at the Faculty of Nursing and Physiotherapy of the University of Alcalá. The study has been approved by the Animal Research and Experimentation Ethics Committee of the University of Alcalá. A total of 60 subjects aged between 18 and 35 with non.specific low back pain will be selected and randomized in two interventions.

The control group will carry out a specific strengthening program for the gluteus maximus and the experimental group will carry out the same strengthening program in addition to receiving a specific manual therapy program for both hips.

The total duration of the treatments will be 8 weeks, with on-treatment evaluations at 4 and 8 weeks, with a follow-up after 1 month.

The objective will be to determine the efficacy of manual therapy on the coxofemoral joint together with a protocol of gluteus maximus strengthening exercises in patients with non-specific chronic low back pain, in comparison with the same protocol of gluteus maximus strengthening exercises performed in isolation, in patients with non-specific chronic low back pain.

DETAILED DESCRIPTION:
Detailed Description has not been entered.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-specific low back pain, with a score of more than 2 on the visual analogue scale.
* Pain with a course of more than 12 weeks, of a chronic nature.

Exclusion Criteria:

* Patients with neurological signs and symptoms or severe psychiatric illnesses.
* Subjects with a history of severe trauma, fracture or previous surgery on the lumbar spine or hip.
* Subjects with a history of musculoskeletal and/or rheumatologic disease.
* Patients with low back pain attributable to dysmenorrhoea.
* Pregnant patients.
* Individuals with fibromyalgia, autoimmune disorders.
* Subjects with a history of oncological processes.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-07-08 (Actual)

PRIMARY OUTCOMES:
Changes in Pain | Baseline, 4 weeks, 8weeks, 1 month after intervention commencement
  measured with visual analogic scale
  A straight horizontal line of fixed length, usually 100 mm is drawn. The ends are defined as the extreme limits of the parameter to be measured (pain) orientated from the left (worst) to the right (best).

SECONDARY OUTCOMES:
Changes in Disability | Baseline, 4 weeks, 8weeks, 1 month after intervention commencement
  measured with the Oswestry Low Back Pain Disability Questionnaire. The interpretation of the scores of this scale varies from 0% to 100%.
  * 0% to 20%: minimal disability: The patient can cope with most living activities.
  * 21%-40%: moderate disability.
  * 41%-60%: severe disability.
  * 61%-80%: crippled.
  * 81%-100%: These patients are either bed-bound or exaggerating their symptoms.
Changes in Health related quality of life | Baseline, 4 weeks, 8weeks, 1 month after intervention commencement
  Using SF-36. This scale is made up of 36 items divided into 8 sections: Physical Function, Function Social, Physical role, Emotional role, Mental health, Vitality, Body pain, General Health. For each of the 8 dimensions, the items are coded, aggregated and transformed into a scale that ranges from 0 (the worst state of health for that dimension) to 100 (the best state of health).
Changes in Depression | Baseline, 4 weeks, 8weeks, 1 month after intervention commencement
  measured with Beck's Depression Inventory
  When the test is scored, a value of 0 to 3 is assigned for each answer and then the total score is compared to a key to determine the depression's severity. The standard cut-off scores were as follows:
  * 0-9: indicates minimal depression
  * 10-18: indicates mild depression
  * 19-29: indicates moderate depression
  * 30-63: indicates severe depression.
  Higher total scores indicate more severe depressive symptoms.
Changes in Gluteus Maximus Strength | Baseline, 4 weeks, 8weeks, 1 month after intervention commencement
  measured with a wireless digital hand-held dynamometer (microFET ® 2). It has a measurement range of 0-300 lbs (pounds). You can select the unit of measurement: pounds, Newtons or Kilogram-force.
  The three main actions of the gluteus maximus will be assessed with respect to its action on the hip: abduction, extension and external rotation.
Changes in the Range of Motion of the Hip Joint | Baseline, 4 weeks, 8weeks, 1 month after intervention commencement
  measured with an 18 cm universal goniometer. The movements to be evaluated are associated with flexion, extension, internal rotation, external rotation, abduction and adduction to end range without pain, explored passively.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Rojas, Principal Investigator — University of Alcalá, Madrid, Spain
Locations (1):
- Manuel Rojas, Madrid, Alcalá de Henares, Spain